CLINICAL TRIAL: NCT04432220
Title: AnticoaguLation ONE Year After Ablation of Atrial Fibrillation in Patients With Atrial Fibrillation (ALONE AF Study)
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2020-0391
Record Dates: First submitted 2020-06-12; First posted 2020-06-16 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Atrial Fibrillation Patients With Moderate or High Stroke Risk Who Had Undergone Catheter Ablation of Atrial Fibrillation
Keywords: catheter ablation; anticoagulation; efficacy; safety

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anticoagulation group(Apixaban group) (Experimental): Apixaban 5mg twice daily (2.5mg twice daily if meets dose-reduction criteria) for 2 years
  Interventions: Drug: Anticoagulation group(Apixaban group)
- Nonanticoagulation group (No Intervention): Standard treatment except anticoagulant for 2 years

INTERVENTIONS:
Drug: Anticoagulation group(Apixaban group) — Apixaban 5mg twice daily (2.5mg twice daily if meets dose-reduction criteria) for 2 years
  Arms: Anticoagulation group(Apixaban group)

SUMMARY:
There has no evidence for the anticoagulation in patients who had undergone catheter ablation of atrial fibrillation, and has maintained sinus rhythm for more than 1 year. However, anticoagulation can increase the risk of bleeding, the study evaluating the role of oral anticoagulation is needed in this patients. This study will compare the efficacy and safety of non-vitamin K anticoagulants (apixaban) and no oral anticoagulation in patient with sinus rhythm one year after catheter ablation of AF.

DETAILED DESCRIPTION:
This study is a prospective randomized study which was performed in multicenter (General Hospital) in Korea. Inclusion criteria is atrial fibrillation patients with moderate or high stroke risk (CHA2DS2-VASc>=1 male, and >=2 female) who had undergone catheter ablation of atrial fibrillation, and has maintained sinus rhythm for more than 1 year. Anticoagulation (Apixaban group) will take apixaban (5 mg bid or 2.5 mg bid according to dose guideline) for 2 years, and nonanticoagulation group will not take any oral anticoagulants for the same period. If the patients have the recurrence of AF, they will take anticoagulation according to standard treatment, and will be censored. We will analyze and compare the efficacy and safety of non-vitamin K anticoagulants (apixaban) and no oral anticoagulation in these patients.

ELIGIBILITY:
Inclusion Criteria:

1. no recurrence of atrial fibrillation one year after catheter ablation of atrial fibrillation
2. CHA2DS2-VASc score >=1 (male) or >=2 (female)
3. age: 19 to 80 years
4. non-valvular atrial fibrillation
5. those who consent the study.
6. those who can be followed after enrollment

Exclusion Criteria:

1. Severe liver or kidney dysfunction
2. Thyroid dysfunction
3. Pregnant or breastfeeding women
4. Malignant tumors that have not been completely cured
5. Severe structural heart disease
6. Predicted survival is less than 12 months
7. Patients who do not understand the content of the study or disagree with it

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — CHA2DS2-VASc score over 1point male or CHA2DS2-VASc score over 2points female.
Enrollment: 840 (Estimated)
Dates: Start 2020-07-28 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Composite outcome | Baseline
  composite outcome including stroke/systemic embolism and major bleeding
Composite outcome | 1 month
  composite outcome including stroke/systemic embolism and major bleeding
Composite outcome | 6 months
  composite outcome including stroke/systemic embolism and major bleeding
Composite outcome | 12 months
  composite outcome including stroke/systemic embolism and major bleeding
Composite outcome | 18 months
  composite outcome including stroke/systemic embolism and major bleeding
Composite outcome | 24 months
  composite outcome including stroke/systemic embolism and major bleeding

SECONDARY OUTCOMES:
Stroke | Baseline
  Ischemic stroke specifically refers to central nervous system infarction (brain, spinal cord, or retinal cell death attributable to ischemia) accompanied by overt symptoms, while silent infarction by definition causes no known symptoms. Stroke also broadly includes intracerebral hemorrhage and subarachnoid hemorrhage.
Stroke | 1 month
  Ischemic stroke specifically refers to central nervous system infarction (brain, spinal cord, or retinal cell death attributable to ischemia) accompanied by overt symptoms, while silent infarction by definition causes no known symptoms. Stroke also broadly includes intracerebral hemorrhage and subarachnoid hemorrhage.
Stroke | 6 months
  Ischemic stroke specifically refers to central nervous system infarction (brain, spinal cord, or retinal cell death attributable to ischemia) accompanied by overt symptoms, while silent infarction by definition causes no known symptoms. Stroke also broadly includes intracerebral hemorrhage and subarachnoid hemorrhage.
Stroke | 12 months
  Ischemic stroke specifically refers to central nervous system infarction (brain, spinal cord, or retinal cell death attributable to ischemia) accompanied by overt symptoms, while silent infarction by definition causes no known symptoms. Stroke also broadly includes intracerebral hemorrhage and subarachnoid hemorrhage.
Stroke | 18 months
  Ischemic stroke specifically refers to central nervous system infarction (brain, spinal cord, or retinal cell death attributable to ischemia) accompanied by overt symptoms, while silent infarction by definition causes no known symptoms. Stroke also broadly includes intracerebral hemorrhage and subarachnoid hemorrhage.
Stroke | 24 months
  Ischemic stroke specifically refers to central nervous system infarction (brain, spinal cord, or retinal cell death attributable to ischemia) accompanied by overt symptoms, while silent infarction by definition causes no known symptoms. Stroke also broadly includes intracerebral hemorrhage and subarachnoid hemorrhage.
Major bleeding | Baseline
  The International Society on Thrombosis and Haemostasis (ISTH)/Scientific and Standardization Committee (SSC) definitions and bleeding assessment tool are useful for standardizing the reporting of bleeding symptoms.
  1. Fatal bleeding. and/or 2. Symptomatic bleeding in a critical area or organ, such as intracranial, intraspinal, intraocular, retroperitoneal, intraarticular or pericardial, or intramuscular with compartment syndrome. and/or 3. Bleeding causing a fall in hemoglobin level of 2 g/dL (1.24 mmol/L) or more, or leading to transfusion of two or more units of whole blood or red cells.
Major bleeding | 1 month
  The International Society on Thrombosis and Haemostasis (ISTH)/Scientific and Standardization Committee (SSC) definitions and bleeding assessment tool are useful for standardizing the reporting of bleeding symptoms.
  1. Fatal bleeding. and/or 2. Symptomatic bleeding in a critical area or organ, such as intracranial, intraspinal, intraocular, retroperitoneal, intraarticular or pericardial, or intramuscular with compartment syndrome. and/or 3. Bleeding causing a fall in hemoglobin level of 2 g/dL (1.24 mmol/L) or more, or leading to transfusion of two or more units of whole blood or red cells.
Major bleeding | 6 months
  The International Society on Thrombosis and Haemostasis (ISTH)/Scientific and Standardization Committee (SSC) definitions and bleeding assessment tool are useful for standardizing the reporting of bleeding symptoms.
  1. Fatal bleeding. and/or 2. Symptomatic bleeding in a critical area or organ, such as intracranial, intraspinal, intraocular, retroperitoneal, intraarticular or pericardial, or intramuscular with compartment syndrome. and/or 3. Bleeding causing a fall in hemoglobin level of 2 g/dL (1.24 mmol/L) or more, or leading to transfusion of two or more units of whole blood or red cells.
Major bleeding | 12 months
  The International Society on Thrombosis and Haemostasis (ISTH)/Scientific and Standardization Committee (SSC) definitions and bleeding assessment tool are useful for standardizing the reporting of bleeding symptoms.
  1. Fatal bleeding. and/or 2. Symptomatic bleeding in a critical area or organ, such as intracranial, intraspinal, intraocular, retroperitoneal, intraarticular or pericardial, or intramuscular with compartment syndrome. and/or 3. Bleeding causing a fall in hemoglobin level of 2 g/dL (1.24 mmol/L) or more, or leading to transfusion of two or more units of whole blood or red cells.
Major bleeding | 18 months
  The International Society on Thrombosis and Haemostasis (ISTH)/Scientific and Standardization Committee (SSC) definitions and bleeding assessment tool are useful for standardizing the reporting of bleeding symptoms.
  1. Fatal bleeding. and/or 2. Symptomatic bleeding in a critical area or organ, such as intracranial, intraspinal, intraocular, retroperitoneal, intraarticular or pericardial, or intramuscular with compartment syndrome. and/or 3. Bleeding causing a fall in hemoglobin level of 2 g/dL (1.24 mmol/L) or more, or leading to transfusion of two or more units of whole blood or red cells.
Major bleeding | 24 months
  The International Society on Thrombosis and Haemostasis (ISTH)/Scientific and Standardization Committee (SSC) definitions and bleeding assessment tool are useful for standardizing the reporting of bleeding symptoms.
  1. Fatal bleeding. and/or 2. Symptomatic bleeding in a critical area or organ, such as intracranial, intraspinal, intraocular, retroperitoneal, intraarticular or pericardial, or intramuscular with compartment syndrome. and/or 3. Bleeding causing a fall in hemoglobin level of 2 g/dL (1.24 mmol/L) or more, or leading to transfusion of two or more units of whole blood or red cells.
Clinically Relivant Non-Major Bleeding (CRNMB) | Baseline, 1month, 6 month, 12 month, 18 month, 24 month
  - Clinically Relivant Non-Major Bleeding (CRNMB) :
  1. Any sign or symptom of hemorrhage (e.g., more bleeding than would be expected for a clinical circumstance, including bleeding found by imaging alone) that does not fit the criteria for the ISTH definition of major bleeding but does meet at least one of the following criteria:
  2. ISTH major bleeding in non-surgical patients is defined as having a symptomatic presentation and 1:
Death | Baseline, 1month, 6 month, 12 month, 18 month, 24 month
  Death: the permanent stopping of all the vital bodily activities
Transient ischemic attack (TIA) | Baseline, 1month, 6 month, 12 month, 18 month, 24 month
  TIA is brief episodes of neurological dysfunction resulting from focal cerebral ischemia not associated with permanent cerebral infarction.
Hospital admission | Baseline, 1month, 6 month, 12 month, 18 month, 24 month
  Hospital admission means admission of a covered person to a hospital as an inpatient for medically necessary and appropriate care and treatment of an Illness or Injury.

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Cardiovascular Hospital Yonsei University, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim D, Shim J, Choi EK, Oh IY, Kim J, Lee YS, Park J, Ko JS, Park KM, Sung JH, Park HW, Park HS, Kim JY, Kang KW, Kim D, Park JK, Kim DH, Kim JB, Yu HT, Kim TH, Uhm JS, Pak HN, Joung B; ALONE-AF Investigators. Long-Term Anticoagulation Discontinuation After Catheter Ablation for Atrial Fibrillation: The ALONE-AF Randomized Clinical Trial. JAMA. 2025 Oct 14;334(14):1246-1254. doi: 10.1001/jama.2025.14679. PMID 40886309